CLINICAL TRIAL: NCT00420550
Title: Pilot Study of Biomarkers and the Relaxation Response Using Guided Imagery in Women With Interstitial Cystitis
Brief Title: Study of Biomarkers and the Relaxation Response Using Guided Imagery in Women With IC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-188
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Interstitial Cystitis; Pelvic Pain
Keywords: Interstitial Cystitis; Pelvic pain; Guided Imagery
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain

INTERVENTIONS:
Behavioral: Relaxation Response using Guided Imagery

SUMMARY:
Interstitial cystitis (IC) affects more than one million women in the United States. It has been thought that IC patients who have been unable to obtain adequate relief from medical remedies would value a psychotherapeutic intervention that could diminish some of their pain.

There are currently no studies using biomarkers with the use of a relaxation technique called guided imagery in IC patients. Many guided imagery intervention studies in areas such as cancer, post-operative pain, and arthritis reported that guided imagery resulted in improvements in the psychological or physiological outcomes examined. If this is also true in IC patients, this intervention may prevent the use of unnecessary medications and procedures that are currently being used.

DETAILED DESCRIPTION:
This is a randomized pilot study. Women who are referred to the Nurse Practitioner for treatment will be invited to enroll. If the patient meets the study criteria, the study will be explained. If the patient agrees to participate in this study, informed consent will be obtained. The patient will be randomized (similar to flipping a coin) into either the Treatment group or Control group. Both groups will be maintained with their IC regimens as prescribed by their own health care providers. The following actions and treatment will done:

There will be 2 visits for all subjects. All subjects will complete a pain diary and medication log during the study. Salivary samples will be obtained at baseline, during the first week of the study, after the 2nd week of the study, the midpoint of the intervention (week 3) and at the end of the study. The Treatment group will listen to a guided imagery CD twice a day, and the Control group will sit or lay down, doing whatever they choose, for the same length of time twice a day. All subjects will complete questionnaires upon enrollment and at week 6.The "Treatment" subjects will receive the guided imagery CD specific for pelvic pain and interstitial cystitis. After the baseline data is completed, they will listen to track 2 of the CD (25 min. in length) twice a day ("Relaxation Exercise A"). The first week they listen to the CD, for 3 days they will obtain salivary tests upon waking then ½ hour later. Then they will listen to the CD, and obtain another salivary sample in addition to recording their pulse and respirations immediately after listening to the CD. The bedtime salivary test, pulse and respirations will be done immediately after listening to the CD. Salivary testing, pulse and respirations will also be done before this evening CD session. The salivary testing will be repeated in the same fashion during the 3rd week of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosed IC patient
* Women at least 18 years of age
* Self reported pelvic pain
* Capable of giving informed consent
* Capable and willing to follow all study related procedures (e.g. keep voiding diary, pain diary, complete questionnaires, listening to CD, obtaining salivary samples).
* Participants must have a stable medication regimen.
* Neuromodulation (if present) must stay stable throughout the study.

Exclusion Criteria:

* Currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function. Patients with neuromodulation devices are excluded for the first 3 months after insertion of the device.
* Use of this guided imagery CD within the past 30 days.
* Diagnosed depression
* Pregnancy or intending to become pregnant during the study
* Cannot independently comprehend and complete the questionnaires.
* The subject is deemed unsuitable for enrollment in this study by the investigators based on their history.
* Men are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Improvement of IC symptoms. Overall improvement will be quantified by a Global Response Assessment.

SECONDARY OUTCOMES:
Bladder symptoms will be assessed by completion of a voiding diary and the Interstitial Cystitis Symptom Index and Problem Index (IC-SIPI) (36) pre- and post- study intervention.
Pain will be measured by a Visual Analog Scale (VAS)
The Relaxation Response will be evaluated by salivary cortisol, alpha amylase and IL-6 levels (all biomarkers), pulse, and respiratory rate.d.) Overall health and well-being will be assessed by the SF-12 (37).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Kusek JW, Nyberg LM. The epidemiology of interstitial cystitis: is it time to expand our definition? Urology. 2001 Jun;57(6 Suppl 1):95-9. doi: 10.1016/s0090-4295(01)01141-4. PMID 11378056
- [Background] Myers DL, Aguilar VC. Gynecologic manifestations of interstitial cystitis. Clin Obstet Gynecol. 2002 Mar;45(1):233-41. doi: 10.1097/00003081-200203000-00024. No abstract available. PMID 11862075